CLINICAL TRIAL: NCT00746499
Title: A Phase 1, Open-Label Study, Investigating First-Dose and Steady-State Pharmacokinetics of Raltegravir in the Genital Tract of HIV Uninfected Women
Brief Title: Pharmacokinetic Study of Raltegravir in Healthy Premenopausal Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IRB #08-0984
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): No control group, only one active arm with subjects taking Raltegravir.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400mg raltegravir BID x 7 days
  Other Names: Isentress

SUMMARY:
Healthy subjects will take study drug by mouth twice a day for 7 consecutive days, blood and cervicovaginal samples will be taken most mornings around the AM dose. Two visits, ~14 hrs in length will be required on Day 1 and 7. The purpose of this study is to measure how much raltegravir is found in the genital tract after taking it orally.

DETAILED DESCRIPTION:
This study is looking at blood and cervicovaginal fluid (CVF) samples of healthy volunteers taking raltegravir. The purpose of this study is to measure the extent that raltegravir penetrates into other body compartments, such as the genital tract. Subjects will take the study drug for 7 days, a total of 10 visits to the research center will be required. A screening visit will occur on no more than 28 days On Days 1 and 7 the subject will stay in the research center for approximately 12 hours for scheduled blood and CVF sampling. Days 3-6 and 8-9 will involve a short visit to the research center for one pre-dose blood and CVF sample before the morning dose. A follow up visit will occur about 7-10 days after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal female subjects
* Between the ages of 18 and 49 years
* With an intact uterus and cervix

(Healthy is defined as no irregular menstrual cycles or clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Negative serum pregnancy test at screening and should be using at least one method of contraception
* Body Mass Index (BMI) of approximately 18 to 30 kg/m^2
* And a total body weight > 50 kg (110 lbs)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Drug levels in CVF and blood plasma | Day 1-9

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States